CLINICAL TRIAL: NCT06500962
Title: SUPeRFOOD: Enhanced SUPport for Initiation and paRticipation in a FOOD is Medicine Program
Brief Title: Enhanced SUPport for Initiation and paRticipation in a FOOD is Medicine Program
Acronym: SUPeRFOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Heart Association (Other); Project Open Hand (Other)
Responsible Party: Principal Investigator, Alexis Beatty, MD, Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 24FIM1259456
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Rehabilitation; Nutrition, Healthy; Nutrition Poor
Keywords: food insecurity; nutrition insecurity; food is medicine
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: 2x2 Factorial Randomization
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (Placebo Comparator)
  Interventions: Behavioral: Usual Care
- Navigation + Usual Care (Experimental)
  Interventions: Behavioral: Usual Care; Behavioral: Navigation
- Text Messaging + Usual Care (Experimental)
  Interventions: Behavioral: Usual Care; Behavioral: Text Messaging
- Navigation + Text Messaging + Usual Care (Experimental)
  Interventions: Behavioral: Usual Care; Behavioral: Navigation; Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Usual Care — Participants will receive a message sent to their electronic health record portal with instructions about how to sign up for a food is medicine program.
Behavioral: Navigation — Participants will receive a weekly phone call from a navigator to promote enrollment in the food is medicine program and address any barriers to participation.
  Arms: Navigation + Text Messaging + Usual Care; Navigation + Usual Care
Behavioral: Text Messaging — Participants will receive two text messages per week to promote healthy eating, enrolling in a food is medicine program, and continuing to participate in a food is medicine program.
  Arms: Navigation + Text Messaging + Usual Care; Text Messaging + Usual Care

SUMMARY:
The purpose of this research is to see if offering more navigation and text-message support will help increase participation and engagement in a Food is Medicine program. The study will recruit people currently participating in cardiac rehabilitation. People will be randomly assigned to 1 of 4 study groups: navigation, text-messaging, both, or neither. People will complete surveys at the start of the study and after 3 months. After 3 months, we will compare how many Food is Medicine meals or groceries people in each group received.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 or older
2. Participating in UCSF Cardiac Rehabilitation
3. Able to communicate in English or Spanish
4. Resident of San Francisco County

Exclusion Criteria

1. Enrolled in hospice
2. Unable to consent for self

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Participant reported satisfaction | 3 months
  Scale of 1 [Quite dissatisfied] to 5 [Very satisfied]

SECONDARY OUTCOMES:
Number of food is medicine meal or grocery distributions received | 3 months
Proportion of participants initiating the food is medicine program | 3 months
  Numerator = number of participants who received at least 1 meal or grocery distribution; Denominator = number of participants in study arm
Proportion of participants engaged in the food is medicine program | 3 months
  Numerator = number of participants who received at least 8 meal or grocery distributions; Denominator = number of participants in study arm

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Dataset and supporting information will be shared on Dryad.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of primary study results

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT06500962/Prot_SAP_000.pdf